CLINICAL TRIAL: NCT03578406
Title: Two-Arm Open-Labeled Trial of HPV-E6-Specific TCR-T Cells With or Without Anti-PD1 Auto-secreted Element in the Treatment of HPV-Positive Head and Neck Carcinoma or Cervical Cancer
Brief Title: HPV-E6-Specific Anti-PD1 TCR-T Cells in the Treatment of HPV-Positive NHSCC or Cervical Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Collaborators: TCRCure Biopharma Ltd. (Industry)
Responsible Party: Principal Investigator, Qingzhu Jia, M.D., Secretary of Research, Xinqiao Hospital of Chongqing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XQDC20180520
Record Dates: First submitted 2018-05-28; First posted 2018-07-06 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cervical Cancer; Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HPV TCR-T (Experimental): HPV E6-specific TCR-T cell
  Interventions: Drug: HPV E6-specific TCR-T cells

INTERVENTIONS:
Drug: HPV E6-specific TCR-T cells — Patients were infused with HPV E6-specific TCR-T cells

SUMMARY:
Human papillomavirus infections 16 (HPV16) is known to be a high-risk factor to induce cervical cancers. To date, HPV16-related cervical cancer is still a major concern in developing countries where vaccination is not prevalent. Concurrent therapies for cervical cancers have limited response rate and high chance of relapse. However, HPV16-induced cancers provided an ideal target for T cell-based immunotherapy due to the non-self origins. Engineered T cells bearing a TCR (TCR-T) that can specifically recognize the presented HPV antigen become a viable approach to treat this type of cancer. Though engineered T therapies have been well-recognized in hematological cancers, solid cancer treatment has been a major hurdle due to the immune-suppressive tumor microenvironment. One key mechanism of tumor-elicited suppression is the PDL1-PD1 interaction which induces T cell exhaustion. Therefore, TCR-T cells armed with a PD1 antagonist could further enhance the efficacy of TCR-T in solid cancers.

ELIGIBILITY:
Inclusion Criteria:

* Expected to live longer than 12 weeks
* PS 0-2
* Pathology confirmed as HPV16 positive malignant tumor, either metastatic or recurrent disease
* Creatinine <2.5mg/dl
* ALT/AST is lower than three times ULN.
* No contraindications of leukocyte collection
* Before entering the trial, women must adopt a reliable method of contraception until 30 days after infusion.
* Understand this trial and have signed an informed consent

Exclusion Criteria:

* Patients with symptomatic brain metastasis
* With other uncontrolled malignant tumors.
* Hepatitis B or Hepatitis C activity period, HIV infected patients
* Any other uncontrolled disease that interferes with the trial
* Patients with severe heart and cerebrovascular diseases such as coronary heart disease, angina pectoris, myocardial infarction, arrhythmia, cerebral thrombosis and cerebral hemorrhage
* Untreated hypertension or hypertensive patients
* A person with a history of mental illness that is difficult to control
* Researchers do not consider it appropriate to participate in this trial
* Patients who have been using immunosuppressive agents for a long time after organ transplants, except for recent or current inhaled corticosteroids
* Subjects who have been pregnant or nursing, or who plan for pregnancy within 2 months of treatment or after the end of treatment
* An illness affects a person who signs a written consent or complies with a study procedure, or who is unwilling or unable to comply with the research requirements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
To Determine the Maximum Tolerated Dose | 8 weeks
  Verify the MTD of TCR-T cells for HPV16 E6 antigen for treatment. Nine patients will be enrolled in this project, using a dose-climbing approach, with every three patients as a group. The first group of patients returned to 5x106/kg TCR-T cells, the second group returned to 1x107/kg TCR-T cells, and the third group returned to 5x107/kg TCR-T cells

CONTACTS AND LOCATIONS:
Overall Officials: Bo Zhu, Principal Investigator — Oncology of Department, Xinqiao Hospital
Locations (1):
- Qingzhu Jia, Chongqing, Chongqing Municipality, China